CLINICAL TRIAL: NCT06494332
Title: Effect of Exercise Combined With Stretching Program to Prevent Lateral Epicondylalgia in Handgun Olympic Shooting Athletes: a Randomized Controlled Trial
Brief Title: Prevention of Lateral Epicondylalgia in Handgun Olympic Shooting Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NB01
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Epicondylitis, Lateral
Keywords: Prevention; Epicaondylalgia; Exercise; Stretching
MeSH Terms: conditions — Tennis Elbow; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 3 weekly sessions (12 sessions in total) of approximately 35 minutes each of exercise and stretching.
  Interventions: Other: Exercise and stretching programe
- Control (No Intervention): No intervention.

INTERVENTIONS:
Other: Exercise and stretching programe — It consists in: a serie of mobility exercises, which were used as warp-up; the mobility of the elbow, forearm, wrist and fingers of both upper limbs was worked on; and, exercises were performed to strengthen the muscles of both forearms.
  Arms: Experimental

SUMMARY:
Lateral epicondylalgia is one of the most common pathologies suffered by Olympic gun shooting athletes. In Spain, there is hardly any research carried out in this sport, so there are no injury prevention protocols available. Preventing these injuries would be fundamental to improve the performance of athletes and to be able to continue adding successes to national honors.

It has also been evidenced that if exercise is combined with stretching, the benefits of physical therapy are increased. High-quality studies have stated that it is not necessary for this exercise protocol combined with stretching to be very prolonged over time, as they affirm that significant improvements can be achieved with only four weeks of exercise.

This study aimed to test the hypothesis that Olympic handgun shooting athletes who perform a four-week multimodal exercise program combined with stretching have a lower risk of suffering from lateral epicondylalgia than athletes who do not perform this program, determining its effectiveness for pain prevention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >35 years
* Present a risk of suffering from lateral epicondylalgia
* Be in possession of a federation Olympic shooting license
* Practice Olympic shooting with handgun and carry out at least one Olympic shooting training session a week or have participated in the last three months in an official competition

Exclusion Criteria:

* Subjects who had serious uncontrolled illnesses
* Who had undergone surgery as a treatment for lateral epicondylalgia
* Who had received treatment for lateral epicondylalgia in the last month or injections of corticosteroids or steroids for this pathology in the last 6 months
* Who had suffered a serious upper limb injury in the last year or present a risk of suffering epicondylalgia due to a cause other than Olympic shooting

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pain - Algometer | 0 week, 4 week
  The algometer will be placed on the lateral epicondyle of the humerus and pressure will be applied until the athlete reported feeling pain. 3 measurements will be made on each upper limb and the average will be obtained.
Pain - Visual Analogic Scale | 0 week, 4 week
  The patients will be shown the Visual Analogic Scale (VAS) scale (0-10) on a sheet of paper and will asked to write down how much pain they had in the lateral epicondyle of each upper limb.

SECONDARY OUTCOMES:
Hand grip strength | 0 week, 4 week
  It will be measured using a manual dynamometer, making 3 measurements on each upper limb with the elbow in flexion and 3 measurements with the elbow in extension, and the average of both methods of measurement will be obtained with the aim of achieving the greatest validity.
Range of movement | 0 week, 4 week
  The active range of elbow joint mobility will be measured by goniometry by a highly experienced researcher. The axis of the goniometer will be placed in the elbow joint, the stationary arm will be placed following the humeral diaphysis and the moving arm will be placed following the diaphysis of the radius. 3 measurements will be made on each upper limb and the average will be obtained in order to achieve the greatest validity.
Subjective perception | 0 week, 4 week
  To assess these subjective variables that can affect sporting performance, a questionnaire has been created with responses using a Likert-type scale from 1 to 5 in which the sensation of stopping and the movement of the handgun is assessed, which are essential elements for the execution of a good shot. Specifically, the aspects analyzed in this questionnaire were the perception of stability when raising the weapon, the perception of the arc of movement when aiming, stopping in the correct area and the sensation of wrist lock when stopping.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Principal Investigator — University of Valencia
Locations (1):
- David Hernández Guillén, Valencia, Spain